CLINICAL TRIAL: NCT04457804
Title: A Brief Virtual ACT Workshop for Emotional Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Barbel Knauper, James McGill Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2020-06-22; First posted 2020-07-07 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Emotional Eating; Eating Behavior
MeSH Terms: conditions — Emotional Eating; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: All participants will be assigned to the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online ACT workshop for Emotional Eating (Experimental): All participants will be assigned to 2, 1.5 hour interventions using Acceptance and Commitment Therapy (ACT) techniques to help reduce emotional eating.
  Interventions: Behavioral: Virtual ACT Workshop for Emotional Eating

INTERVENTIONS:
Behavioral: Virtual ACT Workshop for Emotional Eating — This is a brief online intervention using Acceptance and Commitment Therapy (ACT) technique to target and reduce emotional eating. The intervention will be modeled after Frayn and Knäuper's 1-day ACT workshop for emotional eating intervention, which was derived from Forman and colleagues' "Mind Your Health Program". During the workshop, the following topics will be discussed, based on the three processes of ACT: (1) values clarification/commitment, (2) acceptance/distress tolerance, and (3) mindfulness/awareness.

SUMMARY:
Emotional eating is a behaviour that has been linked to weight concerns, mental health concerns, and disordered eating. Effective interventions have been developed to treat emotional eating, however these exist solely in the context of promoting weight loss. Emotional eating is not exclusive to those who struggle with weight and thus interventions are needed that target those who engage in emotional eating regardless of their weight status. The present study aims to do so through the implementation of a brief online Acceptance and Commitment Therapy (ACT) workshop for emotional eaters.

DETAILED DESCRIPTION:
Emotional eating is defined as increased food consumption in response to negative emotions, and has been linked to weight concerns, mental health concerns, and disordered eating behaviours. Effective interventions have been developed that address emotional eating, namely to improve weight loss. Such interventions are based in Acceptance and Commitment Therapy (ACT), which encourages tolerance of internal cues, such as emotions, and external cues, such as food.

Previous studies have found that brief ACT interventions are effective for the reduction of emotional eating. Our laboratory has recently developed and pilot-tested a one-day ACT workshop intervention for emotional eating, which was found to be effective for reducing emotional eating and deemed feasible and acceptable by participants.

The present study was developed with the aim to adapt the above mentioned workshop intervention to an online format in the context of the COVID-19 crisis. The study aims to test the efficacy, feasibility and acceptability of a brief, online version of the above mentioned one-day ACT workshop for emotional eating. The workshops will be delivered through the Zoom online platform.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifying as emotional-eater
* Being over the age of 18

Exclusion Criteria:

- N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Emotional Eating - Post-Intervention | Assessed at post-intervention (1 week following the first session)
  Emotional eating, as assessed by the Dutch Eating Behaviour Questionnaire Emotional Eating Subscale (DEBQ-EE). Participants are asked to rate the frequency with which they engage in particular eating behaviours, on a 5-point Likert-type rating scale from never (1) to very often (5), with higher scores reflecting higher emotional eating. Only the emotional eating subscale of the DEBQ will be assessed and is calculated by averaging the 13 items that assess emotional eating.
Emotional Eating - 2 weeks post-intervention | Assessed 2-weeks following the second (last) session
  Emotional eating, as assessed by the Dutch Eating Behaviour Questionnaire Emotional Eating Subscale (DEBQ-EE). Participants are asked to rate the frequency with which they engage in particular eating behaviours, on a 5-point Likert-type rating scale from never (1) to very often (5), with higher scores reflecting higher emotional eating. Only the emotional eating subscale of the DEBQ will be assessed and is calculated by averaging the 13 items that assess emotional eating.
Emotional Eating - 3 months Post-Intervention | Assessed 3-months following the second (last) session
  Emotional eating, as assessed by the Dutch Eating Behaviour Questionnaire Emotional Eating Subscale (DEBQ-EE). Participants are asked to rate the frequency with which they engage in particular eating behaviours, on a 5-point Likert-type rating scale from never (1) to very often (5), with higher scores reflecting higher emotional eating. Only the emotional eating subscale of the DEBQ will be assessed and is calculated by averaging the 13 items that assess emotional eating.

SECONDARY OUTCOMES:
Distress Tolerance - Post-Intervention | Assessed at post-intervention (1 week following the first session)
  Distress tolerance, as assessed by the Distress Tolerance Scale (DTS). Participants are asked to indicate the extent to which they agree with statements aimed at assessing distress tolerance, absorption, appraisal, and regulation from 1 (strongly agree) to 5 (strongly disagree), with lower scores reflecting lower distress tolerance. Subscale scores are derived by calculating the means of the items that make up each subscale. Total score is calculating by averaging the four subscales.
Distress Tolerance - 2-weeks Post-Intervention | Assessed 2-weeks following the second (last) session
  Distress tolerance, as assessed by the Distress Tolerance Scale (DTS). Participants are asked to indicate the extent to which they agree with statements aimed at assessing distress tolerance, absorption, appraisal, and regulation from 1 (strongly agree) to 5 (strongly disagree), with lower scores reflecting lower distress tolerance. Subscale scores are derived by calculating the means of the items that make up each subscale. Total score is calculating by averaging the four subscales.
Distress Tolerance - 3-months Post-Intervention | Assessed 3-months following the second (last) session
  Distress tolerance, as assessed by the Distress Tolerance Scale (DTS). Participants are asked to indicate the extent to which they agree with statements aimed at assessing distress tolerance, absorption, appraisal, and regulation from 1 (strongly agree) to 5 (strongly disagree), with lower scores reflecting lower distress tolerance. Subscale scores are derived by calculating the means of the items that make up each subscale. Total score is calculating by averaging the four subscales.
Food Craving Acceptance and Action - Post-intervention | Assessed at post-intervention (1 week following the first session)
  Food craving acceptance and action, as assessed by the Food Craving Acceptance and Action Questionnaire (FAAQ). Items are rated on a 6-point Likert-type rating scale from 1 (very seldom true) to 6 (always true), with higher scores reflecting higher acceptance. Total score is derived by summing all items. Minimum score is 10 and maximum score is 60.
Food Craving Acceptance and Action - 2-weeks Post-intervention | Assessed 2-weeks following the second (last) session
  Food craving acceptance and action, as assessed by the Food Craving Acceptance and Action Questionnaire (FAAQ). Items are rated on a 6-point Likert-type rating scale from 1 (very seldom true) to 6 (always true), with higher scores reflecting higher acceptance. Total score is derived by summing all items. Minimum score is 10 and maximum score is 60.
Food Craving Acceptance and Action - 3-months Post-intervention | Assessed 3-months following the second (last) session
  Food craving acceptance and action, as assessed by the Food Craving Acceptance and Action Questionnaire (FAAQ). Items are rated on a 6-point Likert-type rating scale from 1 (very seldom true) to 6 (always true), with higher scores reflecting higher acceptance. Total score is derived by summing all items. Minimum score is 10 and maximum score is 60.
Mindful Eating - Post-Intervention | Assessed at post-intervention (1 week following the first session)
  Mindful eating, as assessed by the Mindful Eating Questionnaire (MEQ). It is a 28-item self-report measure that assesses five domains of mindful eating: disinhibition, external cues, awareness, emotional response and distraction. Participants are asked to indicate the extent to which extent they agree with each item from 1 ("never" / "rarely") to 4 ("usually"/ "always"), with higher scores reflecting higher levels of mindful eating. Total score is derived by taking the mean of the five subscales.
Mindful Eating - 2-weeks Post-Intervention | Assessed 2-weeks following the second (last) session
  Mindful eating, as assessed by the Mindful Eating Questionnaire (MEQ). It is a 28-item self-report measure that assesses five domains of mindful eating: disinhibition, external cues, awareness, emotional response and distraction. Participants are asked to indicate the extent to which extent they agree with each item from 1 ("never" / "rarely") to 4 ("usually"/ "always"), with higher scores reflecting higher levels of mindful eating. Total score is derived by taking the mean of the five subscales.
Mindful Eating - 3-months Post-Intervention | Assessed 3-months following the second (last) session
  Mindful eating, as assessed by the Mindful Eating Questionnaire (MEQ). It is a 28-item self-report measure that assesses five domains of mindful eating: disinhibition, external cues, awareness, emotional response and distraction. Participants are asked to indicate the extent to which extent they agree with each item from 1 ("never" / "rarely") to 4 ("usually"/ "always"), with higher scores reflecting higher levels of mindful eating. Total score is derived by taking the mean of the five subscales.
ACT Values Application - Post-intervention | Assessed at post-intervention (1 week following the first session)
  Application of ACT values techniques taught during the workshop, as assessed by items developed by the study's authors. Participants were asked to rate the extent to which they agreed with a number of value-based statements on a scale from 1 (strongly disagree) to 5 (strongly agree). Values score was derived by taking the mean of the items, with higher scores reflecting greater value-consistent eating behaviors.
ACT Values Application - 2-weeks Post-intervention | Assessed 2-weeks following the second (last) session
  Application of ACT values techniques taught during the workshop, as assessed by items developed by the study's authors. Participants were asked to rate the extent to which they agreed with a number of value-based statements on a scale from 1 (strongly disagree) to 5 (strongly agree). Values score was derived by taking the mean of the items, with higher scores reflecting greater value-consistent eating behaviors.
ACT Values Application - 3-months Post-intervention | Assessed 3-months following the second (last) session
  Application of ACT values techniques taught during the workshop, as assessed by items developed by the study's authors. Participants were asked to rate the extent to which they agreed with a number of value-based statements on a scale from 1 (strongly disagree) to 5 (strongly agree). Values score was derived by taking the mean of the items, with higher scores reflecting greater value-consistent eating behaviors.
Emotional Eating Frequency - Post-intervention | Assessed at post-intervention (1 week following the first session)
  As assessed by a self-report item developed by the study's authors. Participants were asked to report the number of times they engaged in emotional eating in the past week.
Emotional Eating Frequency - 2-weeks Post-intervention | Assessed 2-weeks following the second (last) session
  As assessed by a self-report item developed by the study's authors. Participants were asked to report the number of times they engaged in emotional eating in the past week.
Emotional Eating Frequency - 3-months Post-intervention | Assessed 3-months following the second (last) session
  As assessed by a self-report item developed by the study's authors. Participants were asked to report the number of times they engaged in emotional eating in the past week.
Ability to Stop Emotional Eating - Post-intervention | Assessed at post-intervention (1 week following the first session)
  As assessed by a single self-report item developed by the study's authors. Participants were asked to report the number of instances in which they began to engage in emotional eating and were able to stop themselves, on a scale from 1 (none of the time) to 5 (very often).
Ability to Stop Emotional Eating - 2-weeks Post-intervention | Assessed 2-weeks following the second (last) session
  As assessed by a single self-report item developed by the study's authors. Participants were asked to report the number of instances in which they began to engage in emotional eating and were able to stop themselves, on a scale from 1 (none of the time) to 5 (very often).
Ability to Stop Emotional Eating - 3-months Post-intervention | Assessed 3-months following the second (last) session
  As assessed by a single self-report item developed by the study's authors. Participants were asked to report the number of instances in which they began to engage in emotional eating and were able to stop themselves, on a scale from 1 (none of the time) to 5 (very often).
Feasibility Data: Recruitment Rates | Assessed during the recruitment period (i.e. over a period of 2 months)
  Overall number of participants who expressed interest in the workshop over the recruitment period.
Feasibility Data: Workshop Attendance Rates | Assessed during the treatment period: from baseline to post-treatment (i.e. over the course of 1 week).
  Number of participants who received the intervention (i.e. who attended both workshop sessions) out of the number of participants who signed up.
Feasibility Data: Dropout Rates | Assessed from baseline to the 3-month follow-up assessment.
  Number of participants who have dropped out or withdrawn from the study at any time point from baseline assessment to last follow-up assessment. Number of dropouts and withdrawals will be kept track of at each study time-point.
Feasibility Data: Loss-to-Follow-Up Rates | Assessed at the 2-week follow-up time point and the 3-month follow-up time point.
  Number of participants (out of those who have attended the workshop) who have not completed the follow-up questionnaire(s). The number of participants with missing follow-up data will be kept track of at all follow-up time points (post-treatment, 2-week follow-up, and 3-month follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Bärbel Knauper, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

REFERENCES:
- [Background] Forman EM, Butryn ML, Juarascio AS, Bradley LE, Lowe MR, Herbert JD, Shaw JA. The mind your health project: a randomized controlled trial of an innovative behavioral treatment for obesity. Obesity (Silver Spring). 2013 Jun;21(6):1119-26. doi: 10.1002/oby.20169. Epub 2013 May 13. PMID 23666772
- [Background] Geliebter A, Aversa A. Emotional eating in overweight, normal weight, and underweight individuals. Eat Behav. 2003 Jan;3(4):341-7. doi: 10.1016/s1471-0153(02)00100-9. PMID 15000995
- [Background] Hou L, Li F, Wang Y, Ou Z, Xu D, Tan W, Dai M. Association between dietary patterns and coronary heart disease: a meta-analysis of prospective cohort studies. Int J Clin Exp Med. 2015 Jan 15;8(1):781-90. eCollection 2015. PMID 25785058
- [Background] Konttinen H, Mannisto S, Sarlio-Lahteenkorva S, Silventoinen K, Haukkala A. Emotional eating, depressive symptoms and self-reported food consumption. A population-based study. Appetite. 2010 Jun;54(3):473-9. doi: 10.1016/j.appet.2010.01.014. Epub 2010 Feb 4. PMID 20138944
- [Background] Lillis J, Niemeier HM, Thomas JG, Unick J, Ross KM, Leahey TM, Kendra KE, Dorfman L, Wing RR. A randomized trial of an acceptance-based behavioral intervention for weight loss in people with high internal disinhibition. Obesity (Silver Spring). 2016 Dec;24(12):2509-2514. doi: 10.1002/oby.21680. Epub 2016 Nov 2. PMID 27804255
- [Background] Oliver G, Wardle J, Gibson EL. Stress and food choice: a laboratory study. Psychosom Med. 2000 Nov-Dec;62(6):853-65. doi: 10.1097/00006842-200011000-00016. PMID 11139006
- [Background] Frayn M, Khanyari S, Knauper B. A 1-day acceptance and commitment therapy workshop leads to reductions in emotional eating in adults. Eat Weight Disord. 2020 Oct;25(5):1399-1411. doi: 10.1007/s40519-019-00778-6. Epub 2019 Sep 20. PMID 31541426
- [Derived] Di Sante J, Frayn M, Angelescu A, Knauper B. Proof-of-concept testing of a brief virtual ACT workshop for emotional eating. Appetite. 2024 Aug 1;199:107386. doi: 10.1016/j.appet.2024.107386. Epub 2024 Apr 30. PMID 38692511

DOCUMENTS (2):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT04457804/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT04457804/SAP_001.pdf